CLINICAL TRIAL: NCT03310957
Title: Single Arm, Open Label Phase 1b/2 Study of SGN-LIV1A in Combination With Pembrolizumab for First-Line Treatment of Patients With Unresectable Locally-Advanced or Metastatic Triple-Negative Breast Cancer
Brief Title: Safety and Efficacy of SGN-LIV1A Plus Pembrolizumab for Patients With Locally-Advanced or Metastatic Triple-Negative Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGNLVA-002; KEYNOTE 721 (Other: Merck Sharp & Dohme LLC); 2017-002289-35 (EudraCT Number); MK-3475-721 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Triple Negative Breast Neoplasms
Keywords: Breast cancer; Breast carcinoma; Triple negative breast cancer; Locally-advanced breast cancer; Metastatic breast cancer; Tumors, breast; Breast tumors; pembrolizumab; LIV-1 protein, human; Ladiratuzumab vedotin; hLIV22-vcMMAE; Seattle Genetics
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — SGN-LIV1A; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LV + pembrolizumab (Experimental): LV + pembrolizumab
  Interventions: Drug: ladiratuzumab vedotin; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ladiratuzumab vedotin — Given into the vein (IV; intravenously)
  Other Names: LV; SGN-LIV1A
Drug: Pembrolizumab — IV infusion every 3 weeks
  Other Names: KEYTRUDA®

SUMMARY:
This trial studies ladiratuzumab vedotin (LV) with pembrolizumab in patients with triple-negative breast cancer. It will find out what side effects happen when participants get these two drugs. A side effect is anything the drugs do besides treating cancer. Pembrolizumab is a drug that can be used to treat triple-negative breast cancer. The trial will also find out if these drugs work to treat this type of cancer. Participants in this study have metastatic breast cancer. This means the cancer has spread to other parts of the body.

DETAILED DESCRIPTION:
The primary goal of this study is to evaluate the combination of LV, which targets LIV-1- expressing tumor cells, with the checkpoint inhibitor pembrolizumab for patients with unresectable locally-advanced or metastatic triple-negative breast cancer. These two drugs act through distinct and possibly complementary modes of action.

This is a single-arm, open-label, multicenter trial. Patients given LV and pembrolizumab during dose escalation will be monitored for frequency of dose-limiting toxicities to determine a recommended doses for expansion cohorts. In addition to safety measures, objective response rate, progression-free survival, overall survival, and other efficacy outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or locally-advanced, histologically documented TNBC (absence of HER2, ER, and PR expression)

  * Part D only: Tumor tissue PD-L1 Combined Positive Score <10 expression.
* Have not previously received cytotoxic therapy for the treatment of unresectable locally-advanced breast cancer or metastatic breast cancer
* At least 6 months since prior treatment with curative intent and recurrence
* At least 1 tumor 10mm in diameter or greater OR lymph node of at least 15 mm in short axis
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Able to provide biopsy tissue for biomarker analysis
* Meet baseline laboratory data criteria

Exclusion Criteria:

* Prior immune-oncology therapy
* Pre-existing neuropathy of at least Grade 2
* History of carcinomatous meningitis or active central nervous system (CNS) metastases. Patients are eligible if CNS metastases are adequately treated and patients have neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 4 weeks prior to enrollment. Patients must be off corticosteroids.
* Received prior radiotherapy within 2 weeks of start of study treatment or have not adequately recovered from prior radiotherapy
* Active autoimmune disease requiring systemic treatment within the past 2 years
* History of interstitial lung disease
* Current pneumonitis or history of pneumonitis requiring steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zejing Wang, MD, PhD, Study Director — Seagen Inc.; Kristel Apolinario, PharmD, Study Director — Seagen Inc.
Locations (50):
- United States (26):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars Sinai Medical Center / Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Chao Family Comprehensive Cancer Center University of California Irvine, Orange, California
  - University of California Irvine - Newport, Orange, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - The Whittingham Cancer Center / Norwalk Hospital, Norwalk, Connecticut
  - Helen F. Graham Cancer Center / Christiana Care Health Systems, Newark, Delaware
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - AdventHealth Cancer Institute, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Winship Cancer Institute / Emory University School of Medicine, Atlanta, Georgia
  - Ingalls Cancer Care / Ingalls Memorial Hospital, Harvey, Illinois
  - Cardinal Bernardin Cancer Center / Loyola University Medical Center, Maywood, Illinois
  - University of Maryland, Baltimore, Maryland
  - Allina Health Cancer Institute, Minneapolis, Minnesota
  - Saint Luke's Cancer Institute LLC, Kansas City, Missouri
  - Summit Medical Group, Florham Park, New Jersey
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - Weill Cornell Medicine, New York, New York
  - University of Pittsburgh Medical Center (UPMC)/Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Texas Oncology - DFW, Dallas, Texas
  - Texas Oncology - Houston Memorial City, Houston, Texas
  - Texas Oncology - San Antonio Medical Center Northeast, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Fred Hutchinson Cancer Center / Seattle Cancer Care Alliance / University of Washington, Seattle, Washington
- Germany (8):
  - Gynakologisches Zentrum Bonn Friedensplatz, Bonn, Other
  - Marien Hospital Bottrop, Bottrop, Other
  - Stadtisches Klinikum Dessau, Dessau, Other
  - Universitatsklinikum Erlangen, Erlangen, Other
  - Kliniken Essen-Mitte - Evang. Huyssens-Stiftung, Essen, Other
  - Rotkreuzklinikum Munich, Munich, Other
  - Klinikum Rechts der Isar der Technischen Universitaet Muenchen, München, Other
  - Klinikum der Universitat Munchen, München
- South Korea (6):
  - Pusan National University Hospital, Busan, Other
  - CHA Bundang Medical Center, Seongnam, Other
  - Korea Cancer Center Hospital, Seoul, Other
  - Seoul National University Hospital, Seoul, Other
  - Severance Hospital, Yonsei University Health System, Seoul, Other
  - Samsung Medical Center, Seoul, Other
- Spain (10):
  - Complejo Hospitalario Universitario La Coruna, A Coruña, Other
  - Hospital del Mar, Barcelona, Other
  - Hospital Universitari Vall d'Hebron, Barcelona, Other
  - Complejo Hospitalario de Jaen, Jaén, Other
  - L'Institut Catala d'Oncologia, L'Hospitalet de Llobregat, Other
  - MD Anderson Cancer Center - Madrid, Madrid, Other
  - Hospital Ruber Internacional, Madrid, Other
  - Hospital Universitario 12 de Octubre, Madrid, Other
  - HM Centro Integral Oncologico Clara Campal, Madrid, Other
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Other

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 185 participants were enrolled at multiple sites.
Pre-assignment Details: Participants were enrolled into Part A, Part B, Part C, and Part D sequentially.
Groups:
- Part A: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab: Participants received SGN-LIV 2.0 milligram per kilogram (mg/kg) by intravenous (IV) infusion on Day 1 of each 21-day cycle every 3 weeks (Q3WK) given over approximately 30 minutes followed by pembrolizumab 200 mg IV as a 30-minute infusion on Day 1 of each 21-day cycle.
- Part A: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab: Participants received SGN-LIV 2.5 mg/kg by IV infusion on Day 1 of each 21-day cycle (Q3WK) given over approximately 30 minutes followed by Pembrolizumab 200 mg IV as a 30-minute infusion on Day 1 of each 21-day cycle in Part A.
- Part B: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab: Participants received SGN-LIV 2.0 mg/kg by IV infusion on Day 1 of each 21-day cycle Q3WK given over approximately 30 minutes followed by pembrolizumab 200 mg IV as a 30-minute infusion on Day 1 of each 21-day cycle in Part B.
- Part B: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab: Participants received SGN-LIV 2.5 mg/kg by IV infusion on Day 1 of each 21-day cycle (Q3WK) given over approximately 30 minutes followed by Pembrolizumab 200 mg IV as a 30-minute infusion on Day 1 of each 21-day cycle in Part B.
- Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab: Participants received SGN-LIV 1.0 mg/kg on Day 1, Day 8, and Day 15 in every 3-week cycle every week (Q1WK) by IV infusion given over approximately 30 minutes followed by pembrolizumab 200 mg as a 30-minute infusion on Day 1 of each 21-day cycle in Part C.
- Part C: SGN-LIV 1.25 mg/kg (Q1WK) + Pembrolizumab: Participants received 1.25 mg/kg on Day 1, 8 and 15 of every 21-day cycle by IV infusion given over approximately 30 minutes followed by 200 mg Pembrolizumab as a 30-minute infusion on Day 1 of each 21-day cycle in Part C.
- Part D: SGN-LIV 1.5 mg/kg (2Q3WK) + Pembrolizumab: Participants received SGN-LIV 1.5 mg/kg on Day 1 and Day 8 of every 21-day cycle twice every 3 weeks (2Q3WK) by IV infusion given over approximately 30 minutes followed by Pembrolizumab 200 mg as a 30-minute infusion on Day 1 of each 21-day cycle in Part D.
Period: Overall Study
Arm/Group | Part A: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab | Part A: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab | Part B: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab | Part B: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab | Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab | Part C: SGN-LIV 1.25 mg/kg (Q1WK) + Pembrolizumab | Part D: SGN-LIV 1.5 mg/kg (2Q3WK) + Pembrolizumab
Started | 7 | 12 | 26 | 47 | 3 | 53 | 37
Treated | 7 | 12 | 26 | 47 | 3 | 53 | 37
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 12 | 26 | 47 | 3 | 53 | 37
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 5 | 0 | 4 | 3
Not completed — Site Terminated | 0 | 1 | 1 | 1 | 0 | 2 | 8
Not completed — Lost to Follow-up | 1 | 1 | 1 | 4 | 0 | 4 | 2
Not completed — Death | 5 | 8 | 18 | 31 | 1 | 29 | 7
Not completed — Discontinuation per sponsor | 0 | 1 | 2 | 4 | 1 | 9 | 12
Not completed — Discontinuation per protocol amendment 11 | 0 | 0 | 0 | 1 | 0 | 3 | 5
Not completed — Treatment landscape | 0 | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Alanine aminotransferase (ALT) increased | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Elevated Aspartate aminotransferase (AST) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Hospice | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Progressive | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: As pre-specified in the statistical analysis plan (SAP), data was summarized by dose levels. Since Arm A and Arm B share the same dose levels (2.0 mg/kg and 2.5 mg/kg), these dose levels were combined across both arms.
Groups:
- Part A, B: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab: Participants received SGN-LIV 2.0 mg/kg by IV infusion on Day 1 of each 21-day cycle Q3WK given over approximately 30 minutes followed by pembrolizumab 200 mg IV as a 30-minute infusion on Day 1 of each 21-day cycle.
- Part A, B: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab: Participants received SGN-LIV 2.5 mg/kg by IV infusion on Day 1 of each 21-day cycle Q3WK given over approximately 30 minutes followed by Pembrolizumab 200 mg IV as a 30-minute infusion on Day 1 of each 21-day cycle.
- Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab: Participants received SGN-LIV 1.0 mg/kg on Day 1, Day 8, and Day 15 in every 3-week cycle Q1WK by IV infusion given over approximately 30 minutes followed by pembrolizumab 200 mg as a 30-minute infusion on Day 1 of each 21-day cycle.
- Part C: SGN-LIV 1.25 mg/kg (Q1WK) + Pembrolizumab: Participants received 1.25 mg/kg on Day 1, 8 and 15 of every 21-day cycle by IV infusion given over approximately 30 minutes followed by 200 mg Pembrolizumab as a 30-minute infusion on Day 1 of each 21-day cycle.
- Part D: SGN-LIV 1.5 mg/kg (2Q3WK) + Pembrolizumab: Participants received SGN-LIV 1.5 mg/kg on Day 1 and Day 8 of every 21-day cycle 2Q3WK by IV infusion given over approximately 30 minutes followed by Pembrolizumab 200 mg as a 30-minute infusion on Day 1 of each 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | Part A, B: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab | Part A, B: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab | Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab | Part C: SGN-LIV 1.25 mg/kg (Q1WK) + Pembrolizumab | Part D: SGN-LIV 1.5 mg/kg (2Q3WK) + Pembrolizumab | Total
Number analyzed (Participants) | 33 | 59 | 3 | 53 | 37 | 185
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: As pre-specified in the SAP, data was summarized by dose levels. Since Arm A and Arm B share the same dose levels (2.0 mg/kg and 2.5 mg/kg), these dose levels were combined across both arms.
  Years | 53.4 (12.1) | 55.2 (12.7) | 45.0 (14.1) | 57.6 (12.7) | 54.6 (11.0) | 55.4 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: As pre-specified in the SAP, data was summarized by dose levels. Since Arm A and Arm B share the same dose levels (2.0 mg/kg and 2.5 mg/kg), these dose levels were combined across both arms.
  Participants
    Female | 33 | 59 | 3 | 53 | 37 | 185
    Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: As pre-specified in the SAP, data was summarized by dose levels. Since Arm A and Arm B share the same dose levels (2.0 mg/kg and 2.5 mg/kg), these dose levels were combined across both arms.
  Participants
    Hispanic or Latino | 4 | 7 | 0 | 5 | 4 | 20
    Not Hispanic or Latino | 29 | 45 | 2 | 43 | 29 | 148
    Unknown or Not Reported | 0 | 7 | 1 | 5 | 4 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race is reported. Population: As pre-specified in the SAP, data was summarized by dose levels. Since Arm A and Arm B share the same dose levels (2.0 mg/kg and 2.5 mg/kg), these dose levels were combined across both arms.
  Participants
    White | 19 | 44 | 0 | 31 | 33 | 127
    Black or African American | 9 | 8 | 1 | 10 | 3 | 31
    Asian | 4 | 1 | 1 | 6 | 1 | 13
    American Indian or Alaska Native | 0 | 1 | 0 | 2 | 0 | 3
    Unknown | 0 | 5 | 1 | 4 | 0 | 10
    Other | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a study participant administered a medicinal product and which did not necessarily have a causal relationship with the study treatment. SAEs was defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria: death, life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly or birth defect and other medically significant events. TEAEs were defined as newly occurring (not present at baseline) or worsened after first dose of investigational product within 30 days after last dose date or within 90 days for SAE. AEs included SAEs and all non-SAEs.
Time Frame: From start of study treatment up to 30 days and up to 90 days post last dose for AEs and SAEs respectively (maximum exposure to any study treatment = 27 months; follow-up: AEs = maximum up to 28 months; SAEs = maximum up to 30 months)
Population: Safety analysis set included all participants who received any amount of SGN-LIV1A or pembrolizumab. As pre-specified in the SAP, data was summarized by dose levels. Since Arm A and Arm B share the same dose levels (2.0 mg/kg and 2.5 mg/kg), these dose levels were combined across both arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, B: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab | Part A, B: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab | Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab | Part C: SGN-LIV 1.25 mg/kg (Q1WK) + Pembrolizumab | Part D: SGN-LIV 1.5 mg/kg (2Q3WK) + Pembrolizumab
Number analyzed (Participants) | 32 | 59 | 2 | 53 | 36
Participants
  Participants With TEAEs | 32 | 59 | 2 | 53 | 36
  Participants With SAEs | 17 | 35 | 1 | 28 | 14

2. Primary Outcome: Number of Participants With Treatment Related TEAEs and SAEs
Description: An AE was any untoward medical occurrence in a study participant administered a medicinal product and which did not necessarily have a causal relationship with the study treatment. SAEs was defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria: death, life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly or birth defect and other medically significant events. AEs included SAEs and all non-SAEs. A treatment-related AE was any untoward medical occurrence attributed to the study drug in a participant who received study drug. AEs were defined as treatment emergent if they were newly occurring or worsened following study treatment. Relatedness to study drug was assessed by the investigator.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, B: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab | Part A, B: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab | Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab | Part C: SGN-LIV 1.25 mg/kg (Q1WK) + Pembrolizumab | Part D: SGN-LIV 1.5 mg/kg (2Q3WK) + Pembrolizumab
Number analyzed (Participants) | 32 | 59 | 2 | 53 | 36
Participants
  Participants With Treatment Related TEAEs | 29 | 58 | 2 | 52 | 35
  Participants With Treatment Related SAEs | 6 | 20 | 0 | 20 | 8

3. Primary Outcome: Number of Participants With AEs of Grade <3 and Grade >=3 Per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v 4.03
Description: An AE was any untoward medical occurrence in a study participant administered a medicinal product and which did not necessarily have a causal relationship with the study treatment. AEs severities were graded using the NCI CTCAE v4.03; where Grade 1= mild AE, Grade 2= moderate AE, Grade 3= severe AE, and Grade 4= life-threatening consequences; urgent intervention indicated, Grade 5= indicated death related to AE.
Time Frame: From start of study treatment up to 30 days for AEs (maximum exposure to any study treatment = 27 months; follow-up: AEs = maximum up to 28 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, B: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab | Part A, B: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab | Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab | Part C: SGN-LIV 1.25 mg/kg (Q1WK) + Pembrolizumab | Part D: SGN-LIV 1.5 mg/kg (2Q3WK) + Pembrolizumab
Number analyzed (Participants) | 32 | 59 | 2 | 53 | 36
Participants
  < Grade 3 | 10 | 10 | 0 | 6 | 5
  >= Grade 3 | 22 | 49 | 2 | 47 | 31

4. Primary Outcome: Number of Participants With Maximum Post-Baseline Laboratory Toxicity Grade (0 to 4) in Any Hematology Parameter
Description: In this outcome measure, number of participants with maximum post-baseline laboratory toxicity grade in any hematology parameter are reported. As per NCI-CTCAE v4.03: Grade 1= mild, Grade 2= moderate, Grade 3= severe, and Grade 4= life-threatening consequences; urgent intervention indicated; Grade 0 = within normal limits. Baseline was defined as most recent non-missing lab result before first dose. Hematology parameters evaluated: hemoglobin, leukocytes, lymphocytes, neutrophils and platelets.
Time Frame: Post-baseline up to 30 days after last dose (maximum exposure to any study intervention was 27 months; follow-up = maximum up to 28 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, B: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab | Part A, B: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab | Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab | Part C: SGN-LIV 1.25 mg/kg (Q1WK) + Pembrolizumab | Part D: SGN-LIV 1.5 mg/kg (2Q3WK) + Pembrolizumab
Number analyzed (Participants) | 32 | 59 | 2 | 53 | 36
Participants
  Grade 0 | 2 | 3 | 0 | 4 | 2
  Grade 1 | 6 | 8 | 1 | 6 | 6
  Grade 2 | 12 | 27 | 1 | 25 | 12
  Grade 3 | 8 | 15 | 0 | 14 | 13
  Grade 4 | 1 | 5 | 0 | 4 | 3
  Missing | 3 | 1 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Maximum Post-Baseline Laboratory Toxicity Grade (0 to 4) in Any Serum Chemistry Parameter
Description: In this outcome measure, number of participants with maximum post-baseline laboratory toxicity grade in any serum chemistry parameters are reported. As per NCI-CTCAE v4.03: Grade 1= mild, Grade 2= moderate, Grade 3= severe, and Grade 4= life-threatening consequences; urgent intervention indicated; Grade 0 = within normal limits. Baseline was defined as most recent non-missing lab result before first dose. Serum chemistry parameters evaluated: alanine aminotransferase, albumin, alkaline phosphatase, amylase, aspartate aminotransferase, bilirubin, calcium corrected for albumin, calcium- ionized, creatinine, gamma glutamyl transferase, glucose, lipase, phosphate, potassium, sodium and urate. In this outcome measure, only those grades as rows are reported which had at least one participant for at least 1 reporting group.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, B: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab | Part A, B: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab | Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab | Part C: SGN-LIV 1.25 mg/kg (Q1WK) + Pembrolizumab | Part D: SGN-LIV 1.5 mg/kg (2Q3WK) + Pembrolizumab
Number analyzed (Participants) | 32 | 59 | 2 | 53 | 36
Participants
  Grade 1 | 10 | 9 | 1 | 4 | 12
  Grade 2 | 6 | 4 | 1 | 10 | 4
  Garde 3 | 12 | 37 | 0 | 36 | 17
  Grade 4 | 1 | 9 | 0 | 3 | 3
  Missing | 3 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT): Part A and Part C
Description: DLT : hematologic and/or non-hematologic AE specified in protocol that is considered related to SGN-LIV or the combination and cannot be attributed to pembrolizumab alone including: any clinically significant, non-hematologic AE>= Grade 3 according to NCI CTCAE v4.03, Grade 3 febrile neutropenia, Grade 4 thrombocytopenia or Grade 3 thrombocytopenia associated with clinically significant bleeding that required medical intervention, Grade 4 anemia unrelated to underlying disease, discontinuation during Cycle 1 due to treatment-related toxicity/ inability to receive all 3 doses of SGN-LIV (Days 1, 8, and 15) as participant not met dosing criteria (Part C only)prolonged delay (>2 weeks) in initiating Cycle 2 due to treatment-related toxicity and Grade 5 event (death).
Time Frame: Cycle 1 (up to 21 days)
Population: DLT-evaluable (DE) analysis included all treated participants in Part A who either (1) experienced a DLT or (2) received at least 75% of intended SGN-LIV1A and pembrolizumab doses and were followed for the full DLT evaluation period. This outcome measure was planned to be analyzed only in Part A and Part C arms.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab: Participants received SGN-LIV 2.0 milligram per kilogram (mg/kg) by intravenous (IV) infusion on Day 1 of each 21-day cycle every 3 weeks (Q3WK) given over approximately 30 minutes followed by pembrolizumab 200 mg IV as a 30-minute infusion on Day 1 of each 21-day cycle in Part A.
- Part A: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab: Participants received SGN-LIV 2.5 mg/kg by IV infusion on Day 1 of each 21-day cycle (Q3WK) given over approximately 30 minutes followed by Pembrolizumab 200 mg IV as a 30-minute infusion on Day 1 of each 21-day cycle in Part B.
Arm/Group | Part A: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab | Part A: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab | Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab | Part C: SGN-LIV 1.25 mg/kg (Q1WK) + Pembrolizumab
Number analyzed (Participants) | 7 | 12 | 2 | 2
Participants | 0 | 2 | 0 | 0

7. Primary Outcome: ORR as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors (RECIST) Version (v)1.1
Description: ORR was defined as the percentage of participants with confirmed complete response (CR) or partial response (PR) according to RECIST v1.1. CR: disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR: >=30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Kaplan Meier method was used for analysis.
Time Frame: From start of study treatment up to date of confirmed CR or PR (maximum up to 30 months)
Population: All treated analysis set included all participants who received any amount of SGN-LIV1A or pembrolizumab. As pre-specified in the SAP, data was summarized by dose levels. Since Arm A and Arm B share the same dose levels (2.0 mg/kg and 2.5 mg/kg), these dose levels were combined across both arms.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A, B: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab | Part A, B: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab | Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab | Part C: SGN-LIV 1.25 mg/kg (Q1WK) + Pembrolizumab | Part D: SGN-LIV 1.5 mg/kg (2Q3WK) + Pembrolizumab
Number analyzed (Participants) | 32 | 59 | 2 | 53 | 36
Percentage of participants | 34 [18.6 to 53.2] | 41 [28.1 to 54.3] | 50 [1.3 to 98.7] | 47 [33.3 to 61.4] | 39 [23.1 to 56.5]

8. Secondary Outcome: Duration of Response (DOR) Per RECIST v1.1
Description: DOR = time from first documentation of objective response (subsequently confirmed) per investigator to first documentation of disease progression, or death due to any cause, whichever came first. CR: disappearance of all target lesions. Any pathological lymph nodes (reduction in short axis to <10 mm). PR: >=30% decrease in sum of diameters of target lesions, taking reference baseline sum diameters. Progression: at least a 20% increase in sum of diameters of target lesions, reference smallest sum on study (includes baseline sum if that is smallest on study). In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 0.5 cm. Appearance of one or more new lesions. Kaplan-Meier method used for DOR evaluation. DOR was only calculated for subgroup of participants who achieved a confirmed CR or PR.
Time Frame: From the date of first CR or PR until the date of the first documentation of progression or death, or censoring date, whichever came first (maximum up to 30 months)
Population: All treated analysis set: all participants who received any amount of SGN-LIV1A or pembrolizumab. As pre-specified in the SAP, data was summarized by dose levels. Since Arm A and Arm B share the same dose levels (2.0 mg/kg and 2.5 mg/kg), these dose levels were combined across both arms.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A, B: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab | Part A, B: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab | Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab | Part C: SGN-LIV 1.25 mg/kg (Q1WK) + Pembrolizumab | Part D: SGN-LIV 1.5 mg/kg (2Q3WK) + Pembrolizumab
Number analyzed (Participants) | 11 | 24 | 1 | 25 | 14
Months | 4.5 [2.9 to 6.9] | 5.8 [3.1 to 9.9] | 4.2 [NA to NA] — Upper and lower limit of 95%CI could not be estimated due to insufficient number of participants with events. | 4.4 [3.6 to 6.6] | 8.3 [5.7 to NA] — Lower limit of 95%CI could not be estimated due to insufficient number of participants with events.

9. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as percentage of participants with CR, PR, or stable disease (SD) per RECIST v1.1. CR: disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR: >=30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progression, taking as reference the smallest sum diameters while on study. Progression: at least a 20% increase in the sum of diameters of target lesions, taking as reference smallest sum on study (this includes baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 0.5 cm. Appearance of one or more new lesions. Clopper-Pearson method was used for 95% confidence interval.
Time Frame: From start of study treatment up to date of CR or PR or SD (maximum up to 30 months)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A, B: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab | Part A, B: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab | Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab | Part C: SGN-LIV 1.25 mg/kg (Q1WK) + Pembrolizumab | Part D: SGN-LIV 1.5 mg/kg (2Q3WK) + Pembrolizumab
Number analyzed (Participants) | 32 | 59 | 2 | 53 | 36
Percentage of participants | 59 [40.6 to 76.3] | 81 [69.1 to 90.3] | 50 [1.3 to 98.7] | 77 [63.8 to 87.7] | 69 [51.9 to 83.7]

10. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from start of study treatment to first documentation of disease progression based upon the disease assessment per RECISTv1.1 or clinical progression, or to death due to any cause, whichever came first. Progression: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 0.5 cm. The appearance of one or more new lesions. Kaplan-Meier method was used for PFS evaluation.
Time Frame: From start of study treatment until the date of the first documentation of progression or death, or censoring date, whichever came first (maximum up to 30 months)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A, B: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab | Part A, B: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab | Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab | Part C: SGN-LIV 1.25 mg/kg (Q1WK) + Pembrolizumab | Part D: SGN-LIV 1.5 mg/kg (2Q3WK) + Pembrolizumab
Number analyzed (Participants) | 32 | 59 | 2 | 53 | 36
Months | 3.5 [1.7 to 4.1] | 4.2 [3.9 to 5.6] | 3.3 [1.0 to NA] — Upper limit of 95%CI could not be estimated due to insufficient participants with events. | 4.8 [4.1 to 5.6] | 4.2 [2.7 to 8.3]

11. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from start of study treatment to date of death due to any cause. In the absence of confirmation of death, OS was censored at the last date the participant was known to be alive. Kaplan-Meier method was used for OS evaluation.
Time Frame: From start of study treatment until the date of death, or censoring date, whichever came first (maximum up to 30 months)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A, B: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab | Part A, B: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab | Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab | Part C: SGN-LIV 1.25 mg/kg (Q1WK) + Pembrolizumab | Part D: SGN-LIV 1.5 mg/kg (2Q3WK) + Pembrolizumab
Number analyzed (Participants) | 32 | 59 | 2 | 53 | 36
Months | 14.6 [8.1 to 26.6] | 14.8 [11.9 to 25.9] | NA [NA to NA] — Median and upper -lower limit of 95%CI could not be estimated due to insufficient number of participants with events. Only 1 participant had event with OS of 3.4 months. | 19.4 [11.1 to NA] — Upper limit of 95%CI could not be estimated due to insufficient number of participants with events. | NA [NA to NA] — Median and upper and lower limit of 95%CI could not be estimated due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: From start of study treatment up to 30 days and up to 90 days post last dose for AEs and SAEs respectively (maximum exposure to any study treatment = 27 months; follow-up: AEs = maximum up to 28 months; All-cause mortality, SAEs = maximum up to 30 months)
Description: Same event may appear as both SAE and non-SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE.
Groups:
- Part A: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab: Participants received SGN-LIV 2.0 mg/kg by IV infusion on Day 1 of each 21-day cycle Q3WK given over approximately 30 minutes followed by pembrolizumab 200 mg IV as a 30-minute infusion on Day 1 of each 21-day cycle in Part A.
- Part A: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab: Participants received SGN-LIV 2.5 mg/kg by IV infusion on Day 1 of each 21-day cycle Q3WK given over approximately 30 minutes followed by Pembrolizumab 200 mg IV as a 30-minute infusion on Day 1 of each 21-day cycle in Part A.
- Part B: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab: Participants received SGN-LIV 2.5 mg/kg by IV infusion on Day 1 of each 21-day cycle Q3WK given over approximately 30 minutes followed by Pembrolizumab 200 mg IV as a 30-minute infusion on Day 1 of each 21-day cycle in Part B.
- Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab: Participants received SGN-LIV 1.0 mg/kg on Day 1, Day 8, and Day 15 in every 3-week cycle Q1WK by IV infusion given over approximately 30 minutes followed by pembrolizumab 200 mg as a 30-minute infusion on Day 1 of each 21-day cycle in Part C.
- Part D: SGN-LIV 1.5 mg/kg (2Q3WK) + Pembrolizumab: Participants received SGN-LIV 1.5 mg/kg on Day 1 and Day 8 of every 21-day cycle 2Q3WK by IV infusion given over approximately 30 minutes followed by Pembrolizumab 200 mg as a 30-minute infusion on Day 1 of each 21-day cycle in Part D.
Arm/Group | Part A: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab | Part A: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab | Part B: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab | Part B: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab | Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab | Part C: SGN-LIV 1.25 mg/kg (Q1WK) + Pembrolizumab | Part D: SGN-LIV 1.5 mg/kg (2Q3WK) + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 5/7 | 8/12 | 18/26 | 31/47 | 1/3 | 29/53 | 7/37
Serious Adverse Events (participants affected / at risk) | 4/7 | 8/12 | 13/26 | 27/47 | 1/3 | 28/53 | 14/37
Other Adverse Events (participants affected / at risk) | 7/7 | 12/12 | 23/26 | 47/47 | 2/3 | 53/53 | 36/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab (N=7) | Part A: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab (N=12) | Part B: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab (N=26) | Part B: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab (N=47) | Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab (N=3) | Part C: SGN-LIV 1.25 mg/kg (Q1WK) + Pembrolizumab (N=53) | Part D: SGN-LIV 1.5 mg/kg (2Q3WK) + Pembrolizumab (N=37)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated adverse reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus gastritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymph gland infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute motor-sensory axonal neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brachial plexopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiparaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbosacral plexopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis in device (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab (N=7) | Part A: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab (N=12) | Part B: SGN-LIV 2.0 mg/kg (Q3WK) + Pembrolizumab (N=26) | Part B: SGN-LIV 2.5 mg/kg (Q3WK) + Pembrolizumab (N=47) | Part C: SGN-LIV 1.0 mg/kg (Q1WK) + Pembrolizumab (N=3) | Part C: SGN-LIV 1.25 mg/kg (Q1WK) + Pembrolizumab (N=53) | Part D: SGN-LIV 1.5 mg/kg (2Q3WK) + Pembrolizumab (N=37)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 11 (14) | 0 (0) | 8 (11) | 3 (4)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 5 (9) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (4) | 0 (0) | 13 (21) | 0 (0) | 11 (19) | 11 (26)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (5)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 3 (3) | 2 (2) | 4 (5) | 0 (0) | 3 (3) | 4 (4)
Dry eye (Eye disorders) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 4 (4) | 3 (3)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 3 (3) | 4 (4) | 4 (4) | 0 (0) | 9 (11) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Visual impairment (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (4) | 0 (0) | 3 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 5 (5) | 4 (6) | 11 (12) | 0 (0) | 16 (17) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 7 (9) | 0 (0) | 4 (4) | 4 (5)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3) | 5 (9) | 10 (11) | 21 (25) | 0 (0) | 25 (27) | 12 (14)
Diarrhoea (Gastrointestinal disorders) | 4 (7) | 9 (15) | 5 (7) | 26 (39) | 0 (0) | 30 (44) | 16 (27)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 4 (4) | 0 (0) | 6 (7) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (3) | 1 (1) | 3 (3) | 0 (0) | 6 (7) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (3)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 6 (7) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (9) | 9 (13) | 12 (17) | 32 (38) | 0 (0) | 35 (57) | 20 (22)
Retching (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 4 (4)
Tongue haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (3) | 7 (11) | 4 (6) | 14 (26) | 0 (0) | 17 (33) | 13 (17)
Asthenia (General disorders) | 2 (2) | 3 (5) | 4 (4) | 5 (6) | 0 (0) | 5 (7) | 9 (21)
Catheter site erosion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (6) | 10 (12) | 11 (11) | 31 (35) | 1 (1) | 32 (41) | 16 (17)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2) | 2 (2) | 6 (7) | 0 (0) | 2 (4) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (2) | 2 (2) | 2 (2) | 0 (0) | 6 (9) | 4 (4)
Pain (General disorders) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 1 (1)
Performance status decreased (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 6 (7) | 11 (14) | 0 (0) | 10 (11) | 5 (7)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 3 (3) | 10 (17)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 4 (5) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (2) | 6 (9) | 0 (0) | 6 (13) | 6 (7)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 6 (7) | 2 (2)
Incision site erythema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 4 (4) | 11 (17) | 0 (0) | 19 (24) | 10 (16)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 3 (4) | 10 (19) | 0 (0) | 23 (30) | 11 (16)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 3 (6) | 0 (0) | 2 (3) | 6 (7)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (6) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 3 (3) | 2 (2)
High density lipoprotein decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 9 (10) | 3 (3)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (4) | 2 (2) | 2 (4) | 0 (0) | 4 (4) | 2 (3)
Neutrophil count increased (Investigations) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 6 (7) | 5 (5) | 13 (15) | 1 (1) | 19 (24) | 11 (11)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 7 (8) | 9 (10) | 18 (19) | 0 (0) | 19 (20) | 10 (14)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 7 (9) | 0 (0) | 5 (8) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 10 (11) | 0 (0) | 14 (21) | 10 (11)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (4) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (6) | 7 (10) | 4 (5) | 11 (20) | 0 (0) | 15 (24) | 9 (11)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 5 (6) | 0 (0) | 9 (11) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (6) | 0 (0) | 3 (3) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 4 (4) | 2 (2)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 6 (7) | 8 (9) | 13 (16) | 0 (0) | 14 (20) | 12 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 5 (7) | 4 (5) | 0 (0) | 7 (10) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (7) | 2 (2) | 6 (7) | 0 (0) | 3 (3) | 4 (4)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (3) | 10 (11) | 0 (0) | 7 (7) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (5) | 6 (7) | 4 (4) | 0 (0) | 8 (10) | 6 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 2 (2) | 8 (10) | 0 (0) | 11 (17) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (2) | 3 (5) | 5 (7) | 1 (1) | 14 (18) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 7 (7) | 6 (6)
Headache (Nervous system disorders) | 1 (2) | 5 (5) | 6 (7) | 9 (17) | 0 (0) | 10 (14) | 6 (8)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 5 (5) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 8 (11) | 4 (4)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 5 (7) | 8 (8) | 23 (30) | 0 (0) | 19 (25) | 13 (16)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vocal cord paresis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 7 (8) | 3 (3)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 4 (4) | 5 (6) | 0 (0) | 17 (18) | 6 (6)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 6 (6) | 15 (19) | 0 (0) | 7 (7) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 2 (2) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 5 (5) | 8 (9) | 0 (0) | 6 (7) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (5) | 0 (0) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (7) | 7 (7) | 25 (25) | 1 (1) | 17 (17) | 12 (12)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 5 (5) | 12 (15) | 0 (0) | 13 (13) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 4 (8) | 0 (0) | 5 (7) | 7 (8)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (8) | 5 (5) | 9 (12) | 0 (0) | 7 (7) | 5 (5)
Scab (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 1 (2)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (5) | 3 (4)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 1 (1) | 2 (2) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT03310957/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT03310957/SAP_001.pdf